CLINICAL TRIAL: NCT03821753
Title: The Effect of the Glycemic Variability on Macular Retinal Microcirculation and Cognitive Functions in Patient With Type 1 Diabetes
Acronym: REVADIAB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Délégation de la Recherche Clinique et de l'innovation (DRCI) (Unknown); CRC (Centre de Recherche Clinique) (Unknown); SFD (Société Francophone du Diabète) (Unknown)
Responsible Party: Sponsor
Other Study IDs: K170406J
Record Dates: First submitted 2018-11-26; First posted 2019-01-30 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2018-11

CONDITIONS: Microvascular Complications; Diabetic Retinopathy; Diabetes; Microangiopathy; Angiography
Keywords: Diabetic retinopathy; Glycemic variability; Diabetes; Macular retinal microcirculation; Microangiopathy; Cognitive dysfunction
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with glycemic variability, defined by a coefficient of variation (CV)> 43%, calculated from continuous glucose measurements data by Free Style Libre® (Abbott)
  Interventions: Other: Case
- Control: Patients without glycemic variability, defined by a coefficient of variation (CV) ≤ 43%, calculated from Free Style Libre® data and matched to patients in the Case group for HbA1c (+/- 0.5%)
  Interventions: Other: Control

INTERVENTIONS:
Other: Case — * OCT
  * OCT-Angiography,
  * Retinophotography
  * Neuropsychological tests
  Groups: Case
Other: Control — * OCT
  * OCT-Angiography,
  * Retinophotography
  * Neuropsychological tests
  Groups: Control

SUMMARY:
Revadiab is case-control study aimed to demonstrate that retinal capillary density is altered in patients with type 1 diabetes with glycemic variability compared to those with comparable glycemic control without glycemic variability. An OCT angiography will be used to precisely evaluate retinal capillary density.

A secondary objective will be to evaluate if glycemic variability is associated with cognitive dysfunction, using a neuro psychologic evaluation.

DETAILED DESCRIPTION:
HbA1c doesn't explain all the microvascular complications of diabetes, especially microvascular complications. Glycemic variability is associated with increased oxidative stress, free radicals and endothelial dysfunction; it contributes to the pathogenesis of diabetic complications.

The relationship between glycemic variability and microangiopathic complications especially retinal but also neurological, needs to be studied.

The principal objective of Revadiab study is to demonstrate a correlation between glycemic variability and macular retinal microcirculation in patient with type 1 diabetes.

The secondary objective is to search a correlation between glycemic variability and :

* Alteration of cognitive functions.
* Severity of peripheral diabetic retinopathy and retinal neuronal damage.
* Other micro and macro angiopathic complications.
* Oxidative stress and inflammation.

Two groups of type 1 diabetic patients will be compared:

* Case: Patient with significant glycemic variability.
* Control: Patients without glycemic variability.

The severity of diabetic retinopathy will be evaluated by the degree of occlusion of small vessels in the central retinal region as measured by OCT angiography.

Acts or Product necessary to research :

* Non-invasive retinal imaging (OCT and OCT- Angiography, retinophotography)
* Neuropsychological tests.
* Blood test.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Type 1 diabetes (T1D)
* Using Free FreeStyle
* Diabete evolving for 10 years or more
* Case: Patients with glycemic variability, defined by a coefficient of variation (CV) > 36%, calculated from continuous glucose measurements data by Free Style Libre® (Abbott)
* Controls: Patients without glycemic variability, defined by a coefficient of variation (CV) ≤ 36%, calculated from Free Style Libre® data and matched to patients in the Case group for HbA1c (+/- 0.5%)

Exclusion Criteria:

* Type 2 diabetic patient
* Corticotherapy
* Comorbidity like cancer
* Antecedent of vitreoretinal pathology
* Antecedent of vitreoretinal surgery
* Important cataract, with an important opacity that prevents a reliable evaluation of capillary density in OCT angio
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of adult patients with T1D with more than 10 years of diabetes and users of the FreeStyle Free continuous measurement system.
  Case: Patients with glycemic variability, defined by a coefficient of variation (CV) > 36%, calculated from continuous glucose measurements data by Free Style Libre® (Abbott).
  Controls: Patients without glycemic variability, defined by a coefficient of variation (CV) ≤ 36%, calculated from Free Style Libre® data and matched to patients in the Case group for HbA1c (+/- 0.5%).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Macular capillary density in the external deep capillary network | 3 months
  Macular capillary density in the external deep capillary network measured by OCT-Angiography (no later than 3 months after inclusion)

SECONDARY OUTCOMES:
Macular capillary density in the deep capillary and deep capillary network | 3 months
  Macular capillary density in the deep capillary and deep capillary network measured by OCT-angiography (no later than 3 months after inclusion)
Area of the central avascular zone | 3 months
  Area of the central avascular zone by OCT-Angiography (no later than 3 months after inclusion)
Macular edema presence | 3 months
  Macular edema presence by OCT (no later than 3 months after inclusion)
Layer thickness reduction of the ganglion cells | 3 months
  Layer thickness reduction of the ganglion cells measured by OCT (no later than 3 months after inclusion)
Diabetic retinopathy stage | 3 months
  Diabetic retinopathy stage evaluated with retinographies (no later than 3 months after inclusion)
Development of pre-retinal neovascular vessels and/or pre-papillary | 3 months
  Development of pre-retinal neovascular vessels and/or pre-papillary (no later than 3 months after inclusion)
Occurrence of neovascular complications | 3 months
  Occurrence of neovascular complications: vitreous
Haemorrhage, retina tractional detachment, neovascular glaucoma | 3 months
  Haemorrhage, retina tractional detachment, neovascular glaucoma (no later than 3 months after inclusion)
Renal function evaluation | 3 months
  Renal function evaluation: microalbuminuria and creatinine determination (no later than 3 months after inclusion)
Evaluation of peripheral neuropathy | 3 months
  Evaluation of peripheral neuropathy : monofilament test (no later than 3 months after inclusion)
Ischemic cardiopathy | 3 months
  Measurement method: treatment with angioplasty or coronary artery bypass graft, Assessment of vascular risk by measuring the coronal calcium score, and determination of BNP and troponin. (no later than 3 months after inclusion)
Number of severe hypoglycemia | 3 months
  Number of severe hypoglycemia since 1 year, threshold for hypoglycemia no later than 3 months after inclusion)
Markers of inflammation | 3 months
  characterization of circulating inflammatory and endothelial cells and CRP-US assay
Oxidative stress markers | 3 months
  Oxidative stress markers: Measurements of 8-iso-prostaglandin F2 alpha urinary and 1,5-anhydroglucitol sanguine. (no later than 3 months after inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No